#### University of California, Los Angeles

#### **CONSENT TO PARTICIPATE IN RESEARCH**

Daily Habits and Consumer Preferences Study

Dr. A. Janet Tomiyama, Ph.D. from the Department of Psychology at the University of California, Los Angeles (UCLA) is conducting a research study.

#### Why is this study being done?

The aim of this research is to understand how daily habits affect consumer ratings. For scientific reasons, this consent form does not include complete information about the study hypotheses and the research questions being tested. You will be fully debriefed following your participation in the research.

### What will happen if I take part in this research study?

If you volunteer to participate in this study, the researcher may ask you to do the following:

- In the first lab visit, have your height and weight taken.
- For the next three days/nights after this visit:
  - Wear a wrist device from bedtime to wake up time to measure your sleep.
  - Attach a very small device to your leg to measure physical activity. You can shower and exercise with this device. If it falls off or you take it off, we will provide extra sticky packets. It looks like this:



- Keep track of what you eat using an online food diary.
- In a second lab visit, complete questionnaires about sociodemographics (e.g., gender identity, income), attitudes towards different social groups (e.g., racial minorities, smokers, overweight people), and sleep.
- In this lab visit, provide consumer ratings for different products with and without someone else who has also filled out those questionnaires.
- In this lab visit, rate some food (cookies, chocolate candies, potato chips, and Sprite).
- Do three more days/nights of sleep, physical activity, and eating monitoring.
- In a final lab visit, return the equipment to us and learn more about the study.

### How long will I be in the research study?

In this study, you will visit the lab three times. The first visit will last approximately one hour and a half, the second visit will last one hour, and the last visit will last about half an hour. In between these visits, you will do 3 days of diet, sleep, and physical activity monitoring.

## Are there any potential risks or discomforts that I can expect from this study?

- Potential risks are minimal. There are no known harms or discomforts associated with this study beyond those encountered in normal daily life.
- You may feel uncomfortable answering questions about your attitudes and behaviors. You have the right to skip any questions that make you uncomfortable.
- You may feel uncomfortable interacting with another person who might have different attitudes than you do. You may end your participation at any time.

### Are there any potential benefits if I participate?

You will not directly benefit from your participation in the research.

However, the results of the research may benefit both the field of psychology as well as society, including the contribution to our deepened understanding about how we behave.

### Will I be paid for participating?

You will be paid up to \$225 for your participation: \$25 for each of your three lab visits and \$25 per day for diet, sleep, and activity measurement (6 days total).

# What other choices do I have if I choose not to participate?

If you choose not to participate in this study, you may participate in any other study you wish.

# How will information about me and my participation be kept confidential?

Any information that is obtained in connection with this study and that can identify you will remain confidential. It will be disclosed only with your permission or as required by law. None of your responses will be labeled with your name or any other identifiable information. You will be assigned a random participation code to take the questionnaires, which will not be linked back to you in any way. Likewise, your responses to questionnaires will not and cannot be linked to you or any information that could identify you.

When the study has ended, we will post the data on the Open Science Framework, which is a place where scientists share their data with other scientists and the public. However, this

data will never include any of your personal information and will not include your name or any identifiable information.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents, or samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings. An example would be a court subpoena.

There are some important things that you need to know. The Certificate DOES NOT stop reporting that federal, state or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. The Certificate CANNOT BE USED to stop a sponsoring United States federal or state government agency from checking records or evaluating programs. The Certificate DOES NOT stop disclosures required by the federal Food and Drug Administration (FDA). The Certificate also DOES NOT prevent your information from being used for other research if allowed by federal regulations.

Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about your involvement in this research. It also does not prevent you from having access to your own information.

**How information about you may be used for future research**. Identifiers may be removed and, after such removal, the information could be used for future research studies or distributed to another investigator for future research studies without additional informed consent from the subject or the legally authorized representative.

There are no plans to provide clinically relevant research results to you in this study.

## What are my rights if I take part in this study?

- You can choose whether or not you want to be in this study, and you may withdraw your consent and discontinue participation at any time.
- Whatever decision you make, there will be no penalty to you, and no loss of benefits to which you were otherwise entitled.
- You may refuse to answer any questions that you do not want to answer and still remain in the study.

Who can I contact if I have questions about this study?

The research team:

If you have any questions, comments or concerns about the research, you can talk to the researcher. Please contact:

Dr. A. Janet Tomiyama, Ph.D. 6534 Pritzker Hall 502 Portola Plaza Los Angeles, California 90095 (310) 206-6875 tomiyama@psych.ucla.edu

UCLA Office of the Human Research Protection Program (OHRPP):

If you have questions about your rights as a research subject, or you have concerns or suggestions and you want to talk to someone other than the researchers, you may contact the UCLA OHRPP by phone: (310) 206-2040; by email: participants@research.ucla.edu or by mail: Box 951406, Los Angeles, CA 90095-1406.

You will be given a copy of this information to keep for your records. SIGNATURE OF STUDY PARTICIPANT

| Name of Participant | |
|---------------------------------------|------|
| Signature of Participant | Date |
| SIGNATURE OF PERSON OBTAINING CONSENT | |
| Name of Person Obtaining Consent | |
| Signature of Person Obtaining Consent | Date |